CLINICAL TRIAL: NCT00358150
Title: A Phase 2, Open-Label, Multi-Center Study Evaluating the Efficacy, Safety and Pharmacokinetics of Genz-112638 in Gaucher Type 1 Patients
Brief Title: A Study of the Efficacy and Safety of Eliglustat Tartrate (Genz-112638) in Type 1 Gaucher Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZGD00304; 2005-004732-42 (EudraCT Number); DRI12816 (Other: Sanofi)
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Gaucher Disease, Type 1; Cerebroside Lipidosis Syndrome; Glucocerebrosidase Deficiency Disease; Glucosylceramide Beta-Glucosidase Deficiency Disease; Gaucher Disease, Non-Neuronopathic Form
Keywords: Type 1 Gaucher Disease; Glucocerebrosidase Deficiency Disease
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

ARMS (1):
- Eliglustat tartrate (Experimental)
  Interventions: Drug: Eliglustat tartrate

INTERVENTIONS:
Drug: Eliglustat tartrate — Eliglustat (Genz-112638) capsule as single 50 mg dose on Day 1 then eliglustat 50 mg twice daily (BID) from Day 2 to Day 19, then either eliglustat 50 mg BID (if Genz-99067[active moiety of eliglustat in plasma] trough plasma concentration was greater than or equal to [>=]5 nanogram per milliliter [ng/mL] on Day 10) or eliglustat 100 mg BID(if Genz-99067 trough plasma concentration was less than [<] 5 ng/mL), from day 20 to Year 4. After primary completion date (Week 52) participants underwent treatment interruption period of approximately 2 weeks before continuing same treatment through study completion (Year 9). Participant receiving 100 mg BID could be considered for further dose increase to 150 mg BID at Week 24 if they met certain criteria (for example, had been on treatment for at least 24 months, had not reached therapeutic goals established for participants receiving Cerezyme, and if all other causes for lack of treatment effect had been evaluated and ruled out).
  Other Names: Genz-112638

SUMMARY:
Gaucher disease is a genetic disease that results in a deficiency of an enzyme acid beta-glucosidase, also known as glucocerebrosidase. This enzyme is needed to digest a substrate (lipid) called glucosylceramide and, to a lesser degree, glucosylsphingosine. In participants with Gaucher disease, the liver, spleen, bone marrow and brain show increases in lipid concentration, specifically in cells derived from the monocyte/macrophage system.

Eliglustat tartrate (Genz-112638) is an oral drug that may regulate the Gaucher disease process by decreasing the synthesis of glucosylceramide. The primary objective of this study is to evaluate the efficacy, safety and pharmacokinetics (PK) of eliglustat tartrate, administered as an oral dose of either 50 milligram (mg) twice daily (BID) or 100 mg BID, to men and women with Gaucher disease Type 1 for 52 weeks.

DETAILED DESCRIPTION:
This study consists of several phases: screening (-28 to -1 days), dose adjustment/treatment (Day 1 [treatment baseline] to Day 30), initial steady-state treatment (post-Day 30 through Week 52 post-baseline), a treatment interruption period (Week 52 through approximately Week 54), long-term steady-state treatment (approximately Week 54 through study completion), and safety follow-up (30 to 37 days after a participant withdraws from or completes the study). The Primary Analysis Period is from baseline through Week 52. The Extension Period is from Week 52 through study completion (that is, participant withdrawal, the study is terminated, eliglustat tartrate becomes commercially available, or where applicable, specific regulatory requirements have been met).

ELIGIBILITY:
Inclusion Criteria:

* The participant had a diagnosis of Gaucher Type I disease and a documented deficiency of glucocerebrosidase activity by enzyme assay and was willing and able to provide written informed consent prior to initiating any study-related procedures;
* The participant was 18 to 65 years old and weighed between 50 and 120 kilogram (kg) at enrollment;
* The participant had the following symptoms of Gaucher disease identified within 28 days of enrollment (at screening);

  * Anemia - indicated by hemoglobin measurements taken during the screening phase (8 to 10 gram per deciliter (g/dL) if female, 8 to 11 g/dL if male);
  * Thrombocytopenia - indicated by platelet count measurements taken during the screening phase (60000 to 100000 per cubic millimeter);
  * Splenomegaly, as indicated by magnetic resonance imaging (MRI) or spiral computed tomography (CT) (>= 10 multiples of normal);
* Female participants of child-bearing potential must had a documented negative serum pregnancy test prior to dosing. Female participants agreed to use a reliable method of birth control throughout duration of trial.

Exclusion Criteria:

* Participant had a partial or total splenectomy or infarcted areas of the spleen;
* Participant had documented prior bleeding varices or liver infarction;
* Participant received miglustat within 12 months prior to study enrollment;
* The participant had received an investigational product within 30 days prior to study enrollment;
* Participant had neurologic or pulmonary involvement;
* Participant had new pathological bone involvement or bone crisis in the 12 months prior to enrollment;
* Participant was transfusion-dependent;
* Participant had a documented etiology of anemia due to causes other than Gaucher disease;
* The participant had cardiac functional and/or anatomical abnormalities, a history of cancer or tested positive for human immunodeficiency virus (HIV) antibody or Hepatitis;
* Participant had a clinically significant disease, other than Gaucher disease, including cardiovascular, renal, hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic, or psychiatric disease, other medical conditions, or serious intercurrent illnesses that, in the opinion of the Investigator, might preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-06; Primary Completion 2009-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (17):
- United States (2):
  - New York University, New York, New York
  - New York, New York
- Argentina (6):
  - Aprillus Asistencia e Investigación, Buenos Aires
  - Hospital de Oncologia Maria Curie, Buenos Aires
  - Hospital Ramos Mejia, Buenos Aires
  - IMAI, Buenos Aires
  - Instituto Argentino de Diagnostico y Tratamiento (IADT), Buenos Aires
  - Buenos Aires
- Israel (4):
  - Rambam Medical Center, Haifa
  - Haifa
  - Sha'are Zedek Medical Centre, Jerusalem
  - Jerusalem
- Universita degli Studi di Milano, Milan, Italy
- Mexico (2):
  - Instituto Mexicano del Seguro Social, D.f.
  - Mexico City
- Russia (2):
  - Hematology Research Center of Ministry of Healthcare of the Russian Federation, Moscow
  - Moscow

REFERENCES:
- [Background] McEachern KA, Fung J, Komarnitsky S, Siegel CS, Chuang WL, Hutto E, Shayman JA, Grabowski GA, Aerts JM, Cheng SH, Copeland DP, Marshall J. A specific and potent inhibitor of glucosylceramide synthase for substrate inhibition therapy of Gaucher disease. Mol Genet Metab. 2007 Jul;91(3):259-67. doi: 10.1016/j.ymgme.2007.04.001. Epub 2007 May 16. PMID 17509920
- [Background] Peterschmitt MJ, Burke A, Blankstein L, Smith SE, Puga AC, Kramer WG, Harris JA, Mathews D, Bonate PL. Safety, tolerability, and pharmacokinetics of eliglustat tartrate (Genz-112638) after single doses, multiple doses, and food in healthy volunteers. J Clin Pharmacol. 2011 May;51(5):695-705. doi: 10.1177/0091270010372387. Epub 2010 Sep 23. PMID 20864621
- [Result] Lukina E, Watman N, Arreguin EA, Banikazemi M, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Rosenthal DI, Kaper M, Singh T, Puga AC, Bonate PL, Peterschmitt MJ. A phase 2 study of eliglustat tartrate (Genz-112638), an oral substrate reduction therapy for Gaucher disease type 1. Blood. 2010 Aug 12;116(6):893-9. doi: 10.1182/blood-2010-03-273151. Epub 2010 May 3. PMID 20439622
- [Result] Lukina E, Watman N, Arreguin EA, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Kamath RS, Rosenthal DI, Kaper M, Singh T, Puga AC, Peterschmitt MJ. Improvement in hematological, visceral, and skeletal manifestations of Gaucher disease type 1 with oral eliglustat tartrate (Genz-112638) treatment: 2-year results of a phase 2 study. Blood. 2010 Nov 18;116(20):4095-8. doi: 10.1182/blood-2010-06-293902. Epub 2010 Aug 16. PMID 20713962
- [Result] Kamath RS, Lukina E, Watman N, Dragosky M, Pastores GM, Arreguin EA, Rosenbaum H, Zimran A, Aguzzi R, Puga AC, Norfleet AM, Peterschmitt MJ, Rosenthal DI. Skeletal improvement in patients with Gaucher disease type 1: a phase 2 trial of oral eliglustat. Skeletal Radiol. 2014 Oct;43(10):1353-60. doi: 10.1007/s00256-014-1891-9. Epub 2014 May 10. PMID 24816856
- [Result] Lukina E, Watman N, Dragosky M, Pastores GM, Arreguin EA, Rosenbaum H, Zimran A, Angell J, Ross L, Puga AC, Peterschmitt JM. Eliglustat, an investigational oral therapy for Gaucher disease type 1: Phase 2 trial results after 4 years of treatment. Blood Cells Mol Dis. 2014 Dec;53(4):274-6. doi: 10.1016/j.bcmd.2014.04.002. Epub 2014 May 15. PMID 24835462
- [Derived] Peterschmitt MJ, Foster MC, Ji AJ, Zajdel MB, Cox GF. Plasma glucosylsphingosine correlations with baseline disease burden and response to eliglustat in two clinical trials of previously untreated adults with Gaucher disease type 1. Mol Genet Metab. 2023 Mar;138(3):107527. doi: 10.1016/j.ymgme.2023.107527. Epub 2023 Jan 25. PMID 36739645

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 50 participants were screened of which 24 participants were screen failure. A total of 26 participants were enrolled in this study.
Groups:
- Eliglustat: Eliglustat (Genz-112638) capsule as single 50 milligram (mg) dose on Day 1 then eliglustat 50 mg twice daily (BID) from Day 2 to Day 19, and then either eliglustat 50 mg BID (if Genz-99067 [active moiety of eliglustat in plasma] trough plasma concentration was greater than or equal to [>=] 5 nanogram per milliliter [ng/mL] on Day 10) or eliglustat 100 mg BID (if Genz-99067 trough plasma concentration was less than [<] 5 ng/mL), from day 20 to Year 4. After primary completion date (Week 52) participants underwent treatment interruption period of approximately 2 weeks before continuing the same treatment up to Year 9. Participant receiving 100 mg BID could be considered for a further dose increase to 150 mg BID at Week 24 if they met certain criteria (for example, had been on treatment for at least 24 months, had not reached therapeutic goals established for participants receiving Cerezyme), and if all other causes for lack of treatment effect had been evaluated and ruled out).
Period: Overall Study
Arm/Group | Eliglustat
Started | 26
Completed | 19
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Undefined | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set consists of all participants who signed informed consent and received at least one dose of eliglustat.
Groups:
- Eliglustat: Eliglustat (Genz-112638) capsule as single 50 mg dose on Day 1 then eliglustat 50 mg BID from Day 2 to Day 19, and then either eliglustat 50 mg BID (if Genz-99067 [active moiety of eliglustat in plasma] trough plasma concentration was greater than or equal to [>=] 5 ng/mL on Day 10) or eliglustat 100 mg BID (if Genz-99067 trough plasma concentration was less than [<] 5 ng/mL), from day 20 to Year 4. After primary completion date (Week 52) participants underwent treatment interruption period of approximately 2 weeks before continuing the same treatment up to Year 9. Participant receiving 100 mg BID could be considered for a further dose increase to 150 mg BID at Week 24 if they met certain criteria (for example, had been on treatment for at least 24 months, had not reached therapeutic goals established for participants receiving Cerezyme, and if all other causes for lack of treatment effect had been evaluated and ruled out).
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.47 (12.960)
Gender [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Ashkenazi Jewish | 7
  Non-Jewish Caucasian | 16
  Hispanic | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated as ([weight in kg] divided by [height in cm multiplied by 0.01]^2).
  kilogram per square meter (kg/m^2) | 22.56 (3.529)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 61.47 (11.018)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.12 (9.747)
Hemoglobin [Mean (Standard Deviation); unit: gram per deciliter (g/dL)] | 11.10 (1.674)
Platelet Count [Mean (Standard Deviation); unit: 10^9 cells per liter] | 66.423 (20.1413)
Spleen Volume [Mean (Standard Deviation); unit: Multiples of normal] | 20.04 (12.798)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Demonstrating A Meaningful Clinical Response
Description: A meaningful clinical response was defined as an improvement in at least 2 of the 3 main efficacy parameters: a) an increase in hemoglobin of greater than or equal to (>=) 0.5 gram/deciliter from baseline, b) an increase in platelets of >=15 percent (%) from baseline, c) reduction in total spleen volume of >= 15% from baseline. As hemoglobin, platelets, total spleen volume were abnormal at baseline, within each participant, only those parameters were used in the evaluation of meaningful clinical response which were abnormal at baseline.
Time Frame: Baseline, Year 1
Population: Full analysis set consists of all participants who signed informed consent and received at least one dose of eliglustat.
Measure: Number; unit: percentage of participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percentage of participants | 77

2. Secondary Outcome: Percent Change From Baseline in Spleen Volume at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Percent change in spleen volume = ([spleen volume at specified time points minus spleen volume at baseline] divided by [spleen volume at baseline]) multiplied by 100, where all volumes are in multiples of normal.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: Full analysis set consists of all participants who signed informed consent and received at least one dose of eliglustat. Here 'n' signifies number of participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percent change
  Change at Year 1 (n=22) | -38.5 (11.41)
  Change at Year 2 (n=20) | -52.4 (10.73)
  Change at Year 3 (n=19) | -59.1 (11.68)
  Change at Year 4 (n=18) | -62.5 (11.63)
  Change at Year 5 (n=19) | -63.9 (14.64)
  Change at Year 6 (n=19) | -66.2 (15.72)
  Change at Year 7 (n=19) | -67.8 (15.65)
  Change at Year 8 (n=15) | -67.9 (17.11)
  Change at Year 9 (n=4) | -52.6 (23.97)
  Change at End of Study (n=19) | -68.6 (18.60)

3. Secondary Outcome: Percent Change From Baseline in Liver Volume at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Percent change in liver volume = ([liver volume at specified time points minus liver volume at baseline] divided by [liver volume at baseline]) multiplied by 100, where all volumes are in multiples of normal.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percent change
  Change at Year 1 (n=22) | -16.9 (10.48)
  Change at Year 2 (n=20) | -23.9 (12.81)
  Change at Year 3 (n=19) | -26.8 (12.28)
  Change at Year 4 (n=18) | -28.0 (13.80)
  Change at Year 5 (n=19) | -31.2 (13.90)
  Change at Year 6 (n=19) | -28.4 (23.58)
  Change at Year 7 (n=19) | -36.2 (13.49)
  Change at Year 8 (n=15) | -31.1 (13.51)
  Change at Year 9 (n=4) | -22.0 (18.49)
  Change at End of Study (n=19) | -36.4 (14.91)

4. Secondary Outcome: Absolute Change From Baseline in Hemoglobin at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Absolute change = hemoglobin level at specified time points minus hemoglobin level at baseline.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
g/dL
  Change at Year 1 (n=22) | 1.70 (1.274)
  Change at Year 2 (n=20) | 2.13 (1.507)
  Change at Year 3 (n=18) | 2.47 (1.406)
  Change at Year 4 (n=19) | 2.27 (1.451)
  Change at Year 5 (n=19) | 2.09 (1.746)
  Change at Year 6 (n=18) | 2.01 (1.326)
  Change at Year 7 (n=19) | 2.07 (1.485)
  Change at Year 8 (n=16) | 2.08 (1.748)
  Change at Year 9 (n=4) | 1.00 (1.480)
  Change at End of Study (n=18) | 2.01 (1.785)

5. Secondary Outcome: Percent Change From Baseline in Platelet Count at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Percent change in platelet count = ([platelet count at specified time points minus platelet count at baseline] divided by [platelet count at baseline]) multiplied by 100.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percent change
  Change at Year 1 (n=22) | 41.3 (36.95)
  Change at Year 2 (n=20) | 81.5 (56.01)
  Change at Year 3 (n=18) | 87.9 (65.37)
  Change at Year 4 (n=19) | 95.1 (89.41)
  Change at Year 5 (n=19) | 90.9 (85.42)
  Change at Year 6 (n=17) | 114.3 (102.48)
  Change at Year 7 (n=19) | 99.4 (97.13)
  Change at Year 8 (n=16) | 109.8 (114.73)
  Change at Year 9 (n=3) | 45.4 (56.28)
  Change at End of Study (n=18) | 117.5 (116.91)

6. Secondary Outcome: Percent Change From Baseline in Biomarker (Angiotensin Converting Enzyme) Level at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and End of Study (Up to Year 9)
Population: Full analysis set consists of all participants who signed informed consent and received at least one dose of eliglustat. Here 'n' signifies number of participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percent change
  Change at Year 1 (n=22) | -35.1 (18.87)
  Change at Year 2 (n=20) | -53.5 (21.05)
  Change at Year 3 (n=19) | -56.7 (19.33)
  Change at Year 4 (n=18) | -60.7 (18.44)
  Change at Year 5 (n=19) | -55.7 (22.51)
  Change at Year 6 (n=17) | -61.5 (24.73)
  Change at Year 7 (n=19) | -63.6 (24.64)
  Change at Year 8 (n=16) | -59.2 (21.77)
  Change at Year 9 (n=4) | -55.1 (32.58)
  Change at End of Study (n=18) | -64.7 (23.38)

7. Secondary Outcome: Percent Change From Baseline in Biomarker (Tartrate-Resistant Acid Phosphatase [TRAP]) Level at Year 1 and Year 2
Time Frame: Baseline, Year 1, Year 2
Population: Full analysis set consists of all participants who signed informed consent and received at least one dose of eliglustat. Here 'n' signifies number of participants with available data at specified time points. As per the change in planned analysis, TRAP was not assessed after Year 2.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percent change
  Change at Year 1 (n=22) | -37.0 (11.64)
  Change at Year 2 (n= 10) | -52.5 (10.61)

8. Secondary Outcome: Percent Change From Baseline in Biomarker Chemokine Ligand 18 (CCL18) Level at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and End of Study
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percent change
  Change at Year 1 (n=21) | -49.0 (24.89)
  Change at Year 2 (n=15) | -72.1 (19.11)
  Change at Year 3 (n=18) | -68.6 (17.27)
  Change at Year 4 (n=18) | -80.2 (12.71)
  Change at Year 5 (n=18) | -89.4 (8.48)
  Change at Year 6 (n=18) | -82.7 (11.98)
  Change at Year 7 (n=18) | -78.5 (17.83)
  Change at Year 8 (n=16) | -79.8 (16.19)
  Change at Year 9 (n=4) | -88.6 (6.30)
  Change at End of Study (n=18) | -85.8 (12.92)

9. Secondary Outcome: Percent Change From Baseline in Biomarker (Chitotriosidase) Level at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
percent change
  Change at Year 1 (n=20) | -49.9 (17.17)
  Change at Year 2 (n=18) | -73.5 (14.93)
  Change at Year 3 (n=17) | -76.4 (12.78)
  Change at Year 4 (n=17) | -79.2 (16.18)
  Change at Year 5 (n=17) | -76.7 (19.16)
  Change at Year 6 (n=17) | -74.1 (26.97)
  Change at Year 7 (n=17) | -75.5 (27.88)
  Change at Year 8 (n=14) | -72.5 (29.20)
  Change at Year 9 (n=4) | -61.2 (36.45)
  Change at End of Study (n=17) | -69.8 (36.59)

10. Secondary Outcome: Change From Baseline in 36-Item Short Form (SF-36) Health Survey Scores at Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8 and Year 9 at End of Study
Description: The SF-36 questionnaire, version 2, investigates the participant's health-related quality of life (HRQL). It is a 36-item questionnaire measuring 8 domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting best health-related quality of life. Two summary scale scores were computed from the 8 domain scores: the Physical Component Summary and the Mental Component Summary. Score range for both summary scale ranges from 0 (worst) to 100 (best), with higher scores reflecting best health-related quality of life.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
units on a scale
  Physical Functioning: Change at Year 1 (n=22) | 8.41 (14.670)
  Physical Functioning: Change at Year 2 (n=20) | 9.50 (17.837)
  Physical Functioning: Change at Year 3 (n=17) | 12.65 (18.296)
  Physical Functioning: Change at Year 4 (n=19) | 11.32 (16.231)
  Physical Functioning: Change at Year 5 (n=19) | 10.76 (19.169)
  Physical Functioning: Change at Year 6 (n=19) | 12.63 (17.589)
  Physical Functioning: Change at Year 7 (n=19) | 11.58 (17.955)
  Physical Functioning: Change at Year 8 (n=16) | 11.56 (17.485)
  Physical Functioning: Change at Year 9 (n=4) | 1.25 (2.500)
  Physical Functioning:Change at End of Study (n=19) | 9.28 (17.085)
  Role - Physical: Change at Year 1 (n=22) | 4.55 (22.091)
  Role - Physical: Change at Year 2 (n=20) | 5.31 (27.824)
  Role - Physical: Change at Year 3 (n=17) | 9.56 (24.717)
  Role - Physical: Change at Year 4 (n=19) | 6.58 (26.391)
  Role - Physical: Change at Year 5 (n=19) | 7.57 (28.227)
  Role - Physical: Change at Year 6 (n=19) | 8.88 (25.964)
  Role - Physical: Change at Year 7 (n=19) | 7.89 (25.331)
  Role - Physical: Change at Year 8 (n=16) | 8.59 (29.393)
  Role - Physical: Change at Year 9 (n=4) | -1.56 (18.663)
  Role - Physical: Change at End of Study (n= 19) | 10.53 (24.211)
  Bodily Pain: Change at Year 1 (n= 22) | -0.77 (21.307)
  Bodily Pain: Change at Year 2 (n= 20) | 4.40 (25.050)
  Bodily Pain: Change at Year 3 (n= 17) | 4.24 (21.297)
  Bodily Pain: Change at Year 4 (n= 19) | -2.53 (25.202)
  Bodily Pain: Change at Year 5 (n= 19) | 0.37 (23.104)
  Bodily Pain: Change at Year 6 (n= 19) | -2.32 (26.268)
  Bodily Pain: Change at Year 7 (n= 19) | 1.74 (27.777)
  Bodily Pain: Change at Year 8 (n= 16) | 1.44 (25.532)
  Bodily Pain: Change at Year 9 (n= 4) | 1.00 (19.630)
  Bodily Pain: Change at End of Study (n= 19) | 6.11 (29.603)
  General Health: Change at Year 1 (n= 22) | 10.36 (19.822)
  General Health: Change at Year 2 (n= 20) | 11.30 (24.262)
  General Health: Change at Year 3 (n= 17) | 16.94 (23.485)
  General Health: Change at Year 4 (n= 19) | 15.53 (23.136)
  General Health: Change at Year 5 (n= 19) | 13.58 (23.710)
  General Health: Change at Year 6 (n= 19) | 12.83 (23.443)
  General Health: Change at Year 7 (n= 19) | 15.89 (23.278)
  General Health: Change at Year 8 (n= 16) | 18.19 (20.140)
  General Health: Change at Year 9 (n= 4) | 11.25 (11.087)
  General Health: Change at End of Study (n= 19) | 15.00 (21.422)
  Vitality: Change at Year 1 (n= 22) | 5.68 (17.242)
  Vitality: Change at Year 2 (n= 20) | 7.71 (26.127)
  Vitality: Change at Year 3 (n= 17) | 14.71 (21.188)
  Vitality: Change at Year 4 (n= 19) | 10.20 (20.005)
  Vitality: Change at Year 5 (n= 19) | 13.82 (23.623)
  Vitality: Change at Year 6 (n= 19) | 12.50 (23.936)
  Vitality: Change at Year 7 (n= 19) | 7.57 (22.782)
  Vitality: Change at Year 8 (n= 16) | 15.23 (23.493)
  Vitality: Change at Year 9 (n= 4) | 3.13 (10.825)
  Vitality: Change at End of Study (n= 19) | 15.13 (21.278)
  Social Functioning: Change at Year 1 (n= 22) | -0.57 (23.298)
  Social Functioning: Change at Year 2 (n= 20) | 10.00 (26.470)
  Social Functioning: Change at Year 3 (n= 17) | 9.56 (19.024)
  Social Functioning: Change at Year 4 (n= 19) | 3.29 (25.291)
  Social Functioning: Change at Year 5 (n= 19) | 9.21 (23.140)
  Social Functioning: Change at Year 6 (n= 19) | 9.21 (26.628)
  Social Functioning: Change at Year 7 (n= 19) | 8.55 (20.435)
  Social Functioning: Change at Year 8 (n= 16) | 11.72 (24.778)
  Social Functioning: Change at Year 9 (n= 4) | 3.13 (6.250)
  Social Functioning: Change at End of Study (n= 19) | 9.21 (25.291)
  Role - Emotional: Change at Year 1 (n= 22) | -3.03 (17.733)
  Role - Emotional: Change at Year 2 (n= 20) | 4.58 (20.675)
  Role - Emotional: Change at Year 3 (n= 17) | 2.45 (16.342)
  Role - Emotional: Change at Year 4 (n= 19) | 3.95 (18.916)
  Role - Emotional: Change at Year 5 (n= 19) | 2.19 (22.020)
  Role - Emotional: Change at Year 6 (n= 19) | 3.07 (23.110)
  Role - Emotional: Change at Year 7 (n= 19) | 0.44 (23.485)
  Role - Emotional: Change at Year 8 (n= 16) | 5.21 (19.927)
  Role - Emotional: Change at Year 9 (n= 4) | -10.42 (12.501)
  Role- Emotional: Change at End of study (n= 19) | 1.32 (22.952)
  Mental Health: Change at Year 1 (n= 22) | 0.23 (17.827)
  Mental Health: Change at Year 2 (n= 20) | 1.75 (19.485)
  Mental Health: Change at Year 3 (n=17) | 7.65 (16.117)
  Mental Health: Change at Year 4 (n= 19) | 4.21 (19.809)
  Mental Health: Change at Year 5 (n= 19) | 6.84 (19.945)
  Mental Health: Change at Year 6 (n= 19) | 5.53 (22.785)
  Mental Health: Change at Year 7 (n= 19) | 6.05 (21.186)
  Mental Health: Change at Year 8 (n= 16) | 7.66 (19.989)
  Mental Health: Change at Year 9 (n= 4) | 3.75 (4.787)
  Mental Health: Change at End of Study (n=19) | 8.68 (20.196)
  Physical Component Summary:Change at Year 1(n= 22) | 3.58 (6.263)
  Physical Component Summary:Change at Year 2(n= 20) | 3.81 (7.968)
  Physical Component Summary:Change at Year 3(n= 17) | 5.17 (7.044)
  Physical Component Summary:Change at Year 4(n= 19) | 3.69 (8.195)
  Physical Component Summary:Change at Year 5(n= 19) | 3.75 (8.430)
  Physical Component Summary:Change at Year 6(n= 19) | 3.88 (6.038)
  Physical Component Summary:Change at Year 7(n= 19) | 4.57 (7.892)
  Physical Component Summary:Change at Year 8(n= 16) | 4.36 (6.946)
  Physical Component Summary: Change at Year 9 (n=4) | 1.98 (5.029)
  Physical Component Summary: Change at EOS (n= 19) | 4.70 (7.120)
  Mental Component Summary: Change at Year 1 (n= 22) | -1.03 (8.703)
  Mental Component Summary: Change at Year 2 (n= 20) | 2.04 (10.476)
  Mental Component Summary: Change at Year 3 (n= 17) | 3.45 (7.881)
  Mental Component Summary: Change at Year 4 (n= 19) | 2.11 (10.013)
  Mental Component Summary: Change at Year 5 (n= 19) | 3.50 (10.963)
  Mental Component Summary: Change at Year 6 (n= 19) | 3.03 (12.535)
  Mental Component Summary: Change at Year 7 (n= 19) | 1.94 (10.982)
  Mental Component Summary: Change at Year 8 (n= 16) | 4.59 (10.106)
  Mental Component Summary: Change at Year 9 (n= 4) | -0.52 (1.287)
  Mental Component Summary: Change at EOS (n=19) | 3.73 (11.243)

11. Secondary Outcome: Change From Baseline in Fatigue Severity Scale (FSS) Scores at Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: The FSS is an instrument consisting of 9 self-administered questions that measures the impact of severity of fatigue symptoms on everyday functioning, based on the recall over the past week. Score range for each question ranges from 1 (minimum) to 7 (maximum), where higher score indicates greater severity. FSS total score was calculated by averaging the results of all questions. Total FSS score ranges from 9 (minimum) to 63 (maximum), where higher scores indicates greater severity.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
units on a scale
  Change at Year 1 (n=17) | -0.56 (1.169)
  Change at Year 2 (n=16) | -0.63 (1.388)
  Change at Year 3 (n=14) | -1.37 (1.983)
  Change at Year 4 (n=16) | -1.41 (1.574)
  Change at Year 5 (n=16) | -1.26 (1.418)
  Change at Year 6 (n=15) | -1.21 (1.681)
  Change at Year 7 (n=16) | -0.97 (1.429)
  Change at Year 8 (n=13) | -1.22 (1.489)
  Change at Year 9 (n=4) | -1.20 (1.192)
  Change at End of Study (n=16) | -1.16 (1.665)

12. Secondary Outcome: Number of Participants With Bone Pain Levels During the Past 4 Weeks at Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Bone pain was assessed as a part of Gaucher disease assessment in participants. Participants were categorized as none (no bone pain), very mild bone pain, mild bone pain and moderate bone pain. In this outcome, number of participants with different levels of bone pain at specified time points were reported.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
participants
  None: Baseline (n=26) | 23
  None: Year 1 (n=22) | 17
  None: Year 2 (n=20) | 17
  None: Year 3 (n=19) | 14
  None: Year 4 (n=19) | 14
  None: Year 5 (n=19) | 16
  None: Year 6 (n=19) | 17
  None: Year 7 (n=19) | 15
  None: Year 8 (n=16) | 14
  None: Year 9 (n=4) | 4
  None: End of Study (n=19) | 18
  Very Mild: Baseline (n=26) | 2
  Very Mild: Year 1 (n=22) | 4
  Very Mild: Year 2 (n=20) | 3
  Very Mild: Year 3 (n=19) | 3
  Very Mild: Year 4 (n=19) | 4
  Very Mild: Year 5 (n=19) | 1
  Very Mild: Year 6 (n=19) | 1
  Very Mild: Year 7 (n=19) | 3
  Very Mild: Year 8 (n=16) | 1
  Very Mild: Year 9 (n=4) | 0
  Very Mild: End of Study (n=19) | 1
  Mild: Baseline (n= 26) | 1
  Mild: Year 1 (n= 22) | 1
  Mild: Year 2 (n= 20) | 0
  Mild: Year 3 (n=19) | 2
  Mild: Year 4 (n=19) | 1
  Mild: Year 5 (n=19) | 2
  Mild: Year 6 (n=19) | 1
  Mild: Year 7 (n=19) | 1
  Mild: Year 8 (n=16) | 1
  Mild: Year 9 (n=4) | 0
  Mild: End of Study (n= 19) | 0
  Moderate: Baseline (n=26) | 0
  Moderate: Year 1 (n=22) | 0
  Moderate: Year 2 (n=20) | 0
  Moderate: Year 3 (n=19) | 0
  Moderate: Year 4 (n=19) | 0
  Moderate: Year 5 (n=19) | 0
  Moderate: Year 6 (n=19) | 0
  Moderate: Year 7 (n=19) | 0
  Moderate: Year 8 (n=16) | 0
  Moderate: Year 9 (n=4) | 0
  Moderate: End of Study (n=19) | 0

13. Secondary Outcome: Number of Participants With Mobility Status (MS) at Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Mobillity, i.e. ability to walk was assessed as a part of Gaucher disease assessment in participants.In this outcome, number of participants with their different mobility status (unrestricted mobility, walks with difficulty) at specified time points were reported.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
participants
  MS: Unrestricted Mobility: Baseline (n=26) | 24
  MS: Unrestricted Mobility: Year 1 (n=22) | 22
  MS: Unrestricted Mobility: Year 2 (n=20) | 20
  MS: Unrestricted Mobility: Year 3 (n=19) | 19
  MS: Unrestricted Mobility: Year 4 (n=19) | 19
  MS: Unrestricted Mobility: Year 5 (n=19) | 19
  MS: Unrestricted Mobility: Year 6 (n=19) | 19
  MS: Unrestricted Mobility: Year 7 (n=19) | 19
  MS: Unrestricted Mobility: Year 8 (n=16) | 16
  MS: Unrestricted Mobility: Year 9 (n=4) | 4
  MS: Unrestricted Mobility: End of Study (n=19) | 18
  MS: Walks with Difficulty: Baseline (n=26) | 2
  MS: Walks with Difficulty: Year 1 (n=22) | 0
  MS: Walks with Difficulty: Year 2 (n=20) | 0
  MS: Walks with Difficulty: Year 3 (n=19) | 0
  MS: Walks with Difficulty: Year 4 (n=19) | 0
  MS: Walks with Difficulty: Year 5 (n=19) | 0
  MS: Walks with Difficulty: Year 6 (n=19) | 0
  MS: Walks with Difficulty: Year 7 (n=19) | 0
  MS: Walks with Difficulty: Year 8 (n=16) | 0
  MS: Walks with Difficulty: Year 9 (n=4) | 0
  MS: Walks with Difficulty: End of Study (n=19) | 1

14. Secondary Outcome: Number of Participants With No Bone Crisis at Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Bone crisis was assessed as a part of Gaucher disease assessment in participants. Acute, excruciating episodic bone pain is characteristic of Gaucher bone crisis, which typically causes debilitation lasting several days or longer and requires treatment with immobilization, hydration, and opioid analgesics. Participants were categorized as 0= no bone crisis, 1= 1 bone crisis, and 2= 2 bone crises during the assessment period. In this outcome, number of participants with 0= no bone crises levels at specified time points were reported.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (Up to Year 9)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
participants
  Baseline (n=26) | 26
  Year 1 (n=22) | 22
  Year 2 (n=20) | 20
  Year 3 (n=19) | 19
  Year 4 (n=19) | 19
  Year 5 (n=19) | 19
  Year 6 (n=19) | 19
  Year 7 (n=19) | 19
  Year 8 (n=16) | 16
  Year 9 (n=4) | 4
  End of Study (n=19) | 19

15. Secondary Outcome: Bone Marrow Infiltration: Number of Participants With Improvement From Baseline in Dark Marrow at Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8 and at End of Study (EOS)
Description: Bone marrow infiltration assessments were designed to evaluate improvements in dark marrow using MRI. Each MRI assessment was performed for both femurs and consisted of reviewing 6 different zones (the femoral head, greater trochanter, intertrochanteric region, shaft, distal metaphysis, and condyles). MRI images recorded dark marrow for each zone as either present or not present at baseline. In this outcome, number of participants (for whom dark marrow was present at baseline) with improvement from baseline in dark marrow at each specified time point were reported.
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8 and at End of Study (up to Year 9)
Population: Full analysis set consists of all participants who signed informed consent and received at least one dose of eliglustat. Here 'n' signifies number of participants who were presented with dark marrow at baseline and had data available at specified time points.
Measure: Count of Participants; unit: Participants
Groups:
- Eliglustat: Eliglustat (Genz-112638) capsule as single 50 mg dose on Day 1 then eliglustat 50 mg BID from Day 2 to Day 19, and then either eliglustat 50 mg BID (if Genz-99067 [active moiety of eliglustat in plasma] trough plasma concentration was greater than or equal to [>=] 5 ng/mL on Day 10) or eliglustat 100 mg BID (if Genz-99067 trough plasma concentration was less than [<] 5 ng/mL), from day 20 to Year 4. After primary completion date (Week 52) participants underwent treatment interruption period of approximately 2 weeks before continuing the same treatment up to Year 8. Participant receiving 100 mg BID could be considered for a further dose increase to 150 mg BID at Week 24 if they met certain criteria (for example, had been on treatment for at least 24 months, had not reached therapeutic goals established for participants receiving Cerezyme, and if all other causes for lack of treatment effect had been evaluated and ruled out).
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
Participants
  Femoral Head: Improved: Year 1: (n=16) | 3
  Femoral Head: Improved: Year 2: (n=14) | 2
  Femoral Head: Improved: Year 3: (n=13) | 2
  Femoral Head: Improved: Year 4: (n=13) | 2
  Femoral Head: Improved: Year 5: (n=13) | 4
  Femoral Head: Improved: Year 6: (n=12) | 5
  Femoral Head: Improved: Year 7: (n=13) | 5
  Femoral Head: Improved: Year 8: (n=13) | 5
  Femoral Head: Improved: End of Study: (n=8) | 3
  Greater Trochanter: Improved: Year 1 (n=8) | 3
  Greater Trochanter: Improved: Year 2 (n=7) | 2
  Greater Trochanter: Improved: Year 3 (n=6) | 3
  Greater Trochanter: Improved: Year 4 (n=6) | 3
  Greater Trochanter: Improved: Year 5 (n=7) | 3
  Greater Trochanter: Improved: Year 6 (n=6) | 1
  Greater Trochanter: Improved: Year 7 (n=7) | 1
  Greater Trochanter: Improved: Year 8 (n=7) | 1
  Greater Trochanter: Improved: End of Study (n=4) | 0
  Intertrochanteric Regions: Improved: Year 1 (n=21) | 1
  Intertrochanteric Regions: Improved: Year 2 (n=19) | 3
  Intertrochanteric Regions: Improved: Year 3 (n=18) | 3
  Intertrochanteric Regions: Improved: Year 4 (n=18) | 3
  Intertrochanteric Regions: Improved: Year 5 (n=18) | 5
  Intertrochanteric Regions: Improved: Year 6 (n=17) | 6
  Intertrochanteric Regions: Improved: Year 7 (n=18) | 6
  Intertrochanteric Regions: Improved: Year 8 (n=17) | 7
  Intertrochanteric Regions: Improved: EOS (n=12) | 5
  Shaft: Improved: Year 1 (n= 20) | 1
  Shaft: Improved: Year 2 (n= 18) | 3
  Shaft: Improved: Year 3 (n= 17) | 3
  Shaft: Improved: Year 4 (n= 17) | 3
  Shaft: Improved: Year 5 (n= 17) | 4
  Shaft: Improved: Year 6 (n= 16) | 5
  Shaft: Improved: Year 7 (n= 17) | 5
  Shaft: Improved: Year 8 (n= 16) | 5
  Shaft: Improved: End of Study (n=11) | 4
  Distal Metaphysis: Improved: Year 1 (n=21) | 2
  Distal Metaphysis: Improved: Year 2 (n=19) | 3
  Distal Metaphysis: Improved: Year 3 (n=18) | 4
  Distal Metaphysis: Improved: Year 4 (n=18) | 3
  Distal Metaphysis: Improved: Year 5 (n=18) | 7
  Distal Metaphysis: Improved: Year 6 (n=17) | 8
  Distal Metaphysis: Improved: Year 7 (n=18) | 8
  Distal Metaphysis: Improved: Year 8 (n=17) | 8
  Distal Metaphysis: Improved: End of Study (n=12) | 6
  Condyles: Improved: Year 1 (n=11) | 3
  Condyles: Improved: Year 2 (n=9) | 1
  Condyles: Improved: Year 3 (n=8) | 1
  Condyles: Improved: Year 4 (n=8) | 1
  Condyles: Improved: Year 5 (n=8) | 2
  Condyles: Improved: Year 6 (n=7) | 2
  Condyles: Improved: Year 7 (n=8) | 2
  Condyles: Improved: Year 8 (n=8) | 2
  Condyles: Improved: End of Study (n=5) | 2

16. Secondary Outcome: Lumbar Spine and Femur T-Scores for Bone Mineral Density (BMD) at Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Images of the lumbar spine and femur were obtained by dual energy X-ray absorptiometry (DXA) to determine T-score for each bone area and total bone mineral density. T-scores compares participant's bone density with that of healthy young participant of same gender. The T-score bone density categories were: normal (score >-1), osteopenia (score -2.5 to <=-1), and osteoporosis (score <= -2.5).
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
T-Score
  Lumbar Spine T-Score: Baseline (n= 25) | -1.85 (1.094)
  Lumbar Spine T-Score: Year 1 (n= 20) | -1.43 (1.015)
  Lumbar Spine T-Score: Year 2 (n= 17) | -0.93 (1.268)
  Lumbar Spine T-Score: Year 3 (n= 15) | -1.09 (1.143)
  Lumbar Spine T-Score: Year 4 (n= 15) | -0.88 (1.258)
  Lumbar Spine T-Score: Year 5 (n= 15) | -0.79 (1.116)
  Lumbar Spine T-Score: Year 6 (n= 15) | -0.69 (1.313)
  Lumbar Spine T-Score: Year 7 (n= 15) | -0.59 (1.265)
  Lumbar Spine T-Score: Year 8 (n= 14) | -0.59 (1.294)
  Lumbar Spine T-Score: Year 9 (n= 4) | 0.00 (0.753)
  Lumbar Spine T-Score: End of Study (n= 6) | -0.35 (1.613)
  Femur T-Scores: Baseline (n= 23) | -0.47 (0.894)
  Femur T-Scores: Year 1 (n= 19) | -0.24 (0.954)
  Femur T-Scores: Year 2 (n= 15) | -0.09 (0.991)
  Femur T-Scores: Year 3 (n= 13) | 0.16 (0.987)
  Femur T-Scores: Year 4 (n= 13) | 0.13 (1.044)
  Femur T-Scores: Year 5 (n= 13) | 0.14 (1.016)
  Femur T-Scores: Year 6 (n= 13) | 0.19 (0.946)
  Femur T-Scores: Year 7 (n= 13) | 0.12 (1.021)
  Femur T-Scores: Year 8 (n= 12) | 0.33 (0.907)
  Femur T-Scores: Year 9 (n= 4) | 0.33 (0.618)
  Femur T-Scores: End of Study (n= 6) | 0.18 (1.278)

17. Secondary Outcome: Lumbar Spine and Femur Z-Scores for BMD at Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study
Description: Images of the lumbar spine and femur were obtained by DXA to determine Z-score for each bone area and total bone mineral density. The Z-score bone density categories are: normal (score >-2) and below normal (score <=-2).
Time Frame: Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9 and at End of Study (up to Year 9)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Eliglustat
Number analyzed (Participants) | 26
Z-Score
  Lumbar Spine Z-Score: Baseline (n= 25) | -1.49 (1.055)
  Lumbar Spine Z-Score: Year 1 (n= 20) | -1.11 (0.961)
  Lumbar Spine Z-Score: Year 2 (n= 17) | -0.64 (0.999)
  Lumbar Spine Z-Score: Year 3 (n= 15) | -0.63 (0.984)
  Lumbar Spine Z-Score: Year 4 (n= 15) | -0.48 (1.073)
  Lumbar Spine Z-Score: Year 5 (n= 15) | -0.37 (0.932)
  Lumbar Spine Z-Score: Year 6 (n= 15) | -0.27 (1.100)
  Lumbar Spine Z-Score: Year 7 (n= 15) | -0.14 (1.053)
  Lumbar Spine Z-Score: Year 8 (n= 14) | -0.29 (1.088)
  Lumbar Spine Z-Score: Year 9 (n= 4) | -0.05 (0.885)
  Lumbar Spine Z-Score: End of Study (n= 6) | 0.18 (0.968)
  Femur Z-Scores: Baseline (n= 23) | -0.17 (0.783)
  Femur Z-Scores: Year 1 (n= 19) | 0.04 (0.813)
  Femur Z-Scores: Year 2 (n= 15) | 0.25 (0.787)
  Femur Z-Scores: Year 3 (n= 13) | 0.52 (0.704)
  Femur Z-Scores: Year 4 (n= 13) | 0.48 (0.773)
  Femur Z-Scores: Year 5 (n= 13) | 0.49 (0.741)
  Femur Z-Scores: Year 6 (n= 13) | 0.57 (0.665)
  Femur Z-Scores: Year 7 (n= 13) | 0.52 (0.683)
  Femur Z-Scores: Year 8 (n= 12) | 0.64 (0.693)
  Femur Z-Scores: Year 9 (n= 4) | 0.38 (0.793)
  Femur Z-Scores: End of Study (n= 6) | 0.73 (0.766)

ADVERSE EVENTS:
Time Frame: Up to Year 9.
Description: Safety set: participants who signed informed consent, received at least 1 dose. Data reported as per dose groups (50/100 mg) as well as for all participants. In the event, 1 participant experienced both serious and non-serious forms of same AE, individual was included in numerator (number of participants affected) of each AE table.
Groups:
- Eliglustat 50 mg BID: Participants who received eliglustat capsule as single 50 mg dose on Day 1 followed by eliglustat 50 mg BID from Day 2 to Year 9.
- Eliglustat 100 mg BID: Participants who received eliglustat capsule as single 50 mg dose on Day 1 followed by eliglustat 50 mg capsule BID from Day 2 to Day 19 and then eliglustat 100 mg capsule BID from Day 20 to Year 9.
- Eliglustat: Participants who received eliglustat capsule as a single 50 mg dose on Day 1 then eliglustat 50 mg BID from Day 2 to Day 19, and then either eliglustat 50 mg BID or eliglustat 100 mg BID from Day 20 to Year 9. Participants who discontinued prior to Day 20 dose had their dose group set to missing and are only included in the all participants group. The Eliglustat group contains all participants who were treated with Eliglustat, including 2 participants dosed with 50 mg QD and 1 participant dosed with 150 mg BID for majority of study. Participants who had dose adjustment will be presented in dose group they received for majority of study.
Arm/Group | Eliglustat 50 mg BID | Eliglustat 100 mg BID | Eliglustat
Serious Adverse Events (participants affected / at risk) | 0/5 | 3/18 | 5/26
Other Adverse Events (participants affected / at risk) | 5/5 | 18/18 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat 50 mg BID (N=5) | Eliglustat 100 mg BID (N=18) | Eliglustat (N=26)
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 2 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat 50 mg BID (N=5) | Eliglustat 100 mg BID (N=18) | Eliglustat (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Bone marrow disorder (Blood and lymphatic system disorders) | 2 | 6 | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 1
Left atrial dilatation (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 3
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 2 | 2
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 3 | 3
Pain (General disorders) | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Vessel puncture site swelling (General disorders) | 0 | 1 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 2
Abscess (Infections and infestations) | 0 | 1 | 1
Bacteriuria (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 3 | 3
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 2 | 2
Infected dermal cyst (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 3 | 4
Onychomycosis (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 2 | 3
Tooth infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 5 | 6
Viral infection (Infections and infestations) | 2 | 5 | 7
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Bacterial test positive (Investigations) | 0 | 1 | 1
Blood folate decreased (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 0 | 2 | 2
Body temperature increased (Investigations) | 0 | 2 | 2
Bone density decreased (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Nerve conduction studies abnormal (Investigations) | 1 | 2 | 3
Urinary sediment present (Investigations) | 0 | 1 | 1
Vitamin B12 decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2 | 2
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 4 | 4
Hyperreflexia (Nervous system disorders) | 0 | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 2 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 2
Haematuria (Renal and urinary disorders) | 2 | 2 | 4
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1
Genital pain (Reproductive system and breast disorders) | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 1 | 2
Haematoma (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 2 | 2

LIMITATIONS AND CAVEATS:
Due to the very small number of participants at Year 9, the point estimates of mean and standard deviation are not reliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.